CLINICAL TRIAL: NCT01608698
Title: A Comparison of Body Weight Changing and Side Effects Between Treatment With 30 mcg Ethinylestradiol/2 mg Chlormadinone Acetate (Belara®) and 30 mcg Ethinylestradiol/3 mg Drospirenone (Yasmin®): A Randomized Control Trial
Brief Title: Comparison of Body Weight Change During Contraception With Belara and Yasmin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R015532040; 015532040 (Other Grant/Funding Number: Faculty of Medicine Siriraj Hospital, Mahidol University)
Record Dates: First submitted 2012-05-21; First posted 2012-05-31 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Body Weight Changes
Keywords: chlormadinone acetate; drospirenone; contraceptive pills
MeSH Terms: conditions — Body Weight Changes | interventions — Belara; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belara (Experimental): The participants who receive OCP in combination of 30 mcg ethinylestradiol/2 mg chlormadinone acetate (Belara®).
  Interventions: Drug: 30 mcg ethinylestradiol/2 mg chlormadinone acetate
- Yasmin (Experimental): The participants who receive OCP in combination of 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin®).
  Interventions: Drug: 30 mcg ethinylestradiol/3 mg drospirenone

INTERVENTIONS:
Drug: 30 mcg ethinylestradiol/2 mg chlormadinone acetate — By orally 1 tablet before bedtime for 21 days and withdrawal 7 days after that start the new cycle. Total study period is 6 cycles of pills.
  Other Names: Belara
  Arms: Belara
Drug: 30 mcg ethinylestradiol/3 mg drospirenone — By orally 1 tablet before bedtime for 21 days then withdrawal 7 days after that start the new cycle. Total study period is 6 cycles of pills.
  Other Names: Yasmin
  Arms: Yasmin

SUMMARY:
The purpose of this study is to evaluate different side effect in contraceptive use of two oral combined contraceptive pills (OCP)in combination of 30 mcg ethinylestradiol/2 mg chlormadinone acetate (Belara®) and 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin®), especially body weight change.

DETAILED DESCRIPTION:
Oral combined contraceptive pills (OCP) is the most contraceptive use in reproductive women. The various type of progestins in OCP give various effects either benefit (non-contraceptive benefit) and side effect. These effects depend on pharmacological activity of each progestin. Many studies showed causes of discontinuation use of OCP, such as increase body weight,androgenic effect and vaginal spotting. OCP in combination of 30 mcg ethinylestradiol/2 mg chlormadinone acetate (Belara®) and 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin®)are the common used in practice. The each type of progestin (chlormadinone and drospirenone) might effect different outcomes in women especially in body weight change during use. Chlormadinone is a C-21 progestin which has glucocorticoid and antiandrogenic effect. Drospirenone is a progestin in spironolactone derivative which has antimineralocorticoid and antiandrogenic effect. Both progestins might has less effect in body weight change and provide other non-contraceptive benefits. So investigator want to study the different effects from these progestin in two type of OCP. The result from this study could give information to choose the proper OCP for each reproductive woman.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive woman
* Woman who has BMI < 28.5 kg/m2.
* Woman who has regular menstruation.
* Woman who don't have pelvic organ disorder.
* Woman who want contraception with oral contraceptive pills.

Exclusion Criteria:

* Woman who has abnormal blood pressure
* Woman who has abnormal vaginal bleeding
* Pregnant woman
* Woman who on medication effect contraceptive pills, such as anti-fungal, anti-retroviral, anti-convulsant drug.
* Woman who has contraindication for OCP.
* Woman who use steroid in 3 month period before enrollment in this study.
* Smoking
* Woman who has eating habit disorder.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
body weight change | 6 month
  Compare the body weight change during use of two OCP (30 mcg ethinylestradiol/2 mg chlormadinone acetate (Belara®) and 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin®)). By follow up at 3rd and final at 6th month of use.

SECONDARY OUTCOMES:
efficacy in contraception (pregnancy rate) | 6 month
  To evaluate contraceptive efficacy of two OCP. Urine pregnancy test was used to evaluate pregnancy, the participant was tested in every visit of the study.
Other side effects | 6 month
  To evaluate other side effects during using both OCP,such as vaginal spotting, androgenic effect, blood pressure, headache and GI effect. Vaginal spotting was classified by number of pad (WHO definition) which the participant used in each cycle and record in menstrual card. Androgenic effect was classified by Modified Ferriman - Gallway Score for hirsutism (score > 7), American Academy of Dermatology Consensus 2009 on acne classification (mild, moderate, severe)for acne, systolic/diastolic blood pressure and the presence or no presence of headache and GI discomfort.
satisfaction | 6 month
  To compare satisfaction in study process. In each visit (first, 3rd month and 6th month of study period). The participant was evaluated satisfaction in topics of diagnosis, timing of study process, information from the staff about the study process and the way to use oral pills, quality of the oral pills and conclusive satisfaction. The rating of satisfaction was categorised in five levels as five scoring numbers by using questionnaire; 5=extreme satisfaction, 4=very satisfaction, 3=moderate satisfaction, 2= little satisfaction, 1=no satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Family Planning Unit, Department of Obstetric and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Wongwananuruk T, Panichyawat N, Panchalee T, Jirakittidul P, Angsuwathana S, Sirimai K, Thamkhantho M, Chiravacharadej G. Comparison of change in body weight between contraception containing 30-mug ethinylestradiol/2-mg chlormadinone acetate or 30-mug ethinylestradiol/3-mg drospirenone: a randomised controlled trial. Eur J Contracept Reprod Health Care. 2020 Feb;25(1):43-48. doi: 10.1080/13625187.2019.1688290. Epub 2019 Nov 22. PMID 31756117